CLINICAL TRIAL: NCT02133105
Title: Efficacy of Intravenous Levosimendan Compared With Dobutamine on Renal Hemodynamics and Function in Chronic Heart Failure
Brief Title: Levosimendan Versus Dobutamine for Renal Function in Heart Failure
Acronym: ELDOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-000986-36; 2013-000986-36 (EudraCT Number)
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Cardiorenal Syndrome
Keywords: Heart failure; Renal failure; Inotropic drugs; Levosimendan; Dobutamine
MeSH Terms: conditions — Cardio-Renal Syndrome; Heart Failure; Renal Insufficiency | interventions — Simendan; Dobutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levosimendan (Active Comparator): Levosimendan administration is initiated with a loading dose of 12μg/kg given over 10 min followed by a continuous infusion of 0.1 μg/kg/min for 65 min.
  Interventions: Drug: Levosimendan
- Dobutamine (Active Comparator): Dobutamine is given as a continuous infusion without a bolus dose. The infusion rate is started at 5.0 μg/kg/min for 10 minutes, and thereafter increased to 7,5 μg/kg/min for 65 min.
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Levosimendan
  Other Names: Simdax
  Arms: Levosimendan
Drug: Dobutamine
  Other Names: Dobutrex
  Arms: Dobutamine

SUMMARY:
Although inotropes have a favorable effect on central hemodynamics in patients with heart failure, their effect on renal hemodynamics is incompletely defined. The purpose of this study is to evaluate the efficacy of a 75 min intravenous infusion of levosimendan compared to a 75 min infusion of dobutamine on renal hemodynamics and function in patients with chronic heart failure and signs of cardiorenal syndrome. The investigators hypothesis is that patients treated with levosimendan will show greater increases in renal blood flow and glomerular filtration rate (GFR) than those treated with dobutamine.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed and dated informed consent
* Male and Female subjects ≥18 years of age
* Chronic congestive heart failure scheduled for right sided cardiac catheterization
* Left ventricular ejection fraction ≤ 40% determined by echocardiography
* Elevation of N Terminal-proBNP ≥ 500 ng/L
* Cardiorenal syndrome (30ml/min ≤ estimated GFR ≤ 80 ml/min (MDRD)

Exclusion Criteria:

* Acute heart failure, untreated
* Systolic blood pressure < 80 mmHg
* Tachycardia above 100 bpm
* Angina Canadian Cardiovascular Society (CCS) class III or higher
* Aortic stenosis
* Hypertrophic cardiomyopathy
* Restrictive cardiomyopathy
* The presence of kidney disease diagnosed before heart failure
* Administration of radiographic contrast < 1 week
* Radiographic contrast allergy
* In the Investigator's opinion, the patient has a clinically significant disease that could be adversely affected by study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in renal blood flow | 75 min minus baseline
  Para-aminohippuric acid (PAH) infusion clearance
Change in glomerular filtration rate | 75 min minus baseline
  Chrome-ethylenediaminetetraacetic acid (EDTA) infusion clearance

SECONDARY OUTCOMES:
Change in renal vascular resistance | 75 min minus baseline
  Renal blood flow divided by the difference between renal arterial pressure and renal venous pressure
Change in central hemodynamics | 75 min minus baseline
  Right atrial pressure, mean pulmonary arterial pressure, pulmonary capillary wedge pressure, mean arterial pressure, cardiac output, pulmonary vascular resistance and systemic vascular resistance measured with a pulmonary artery thermodilution catheter.
Change in renal oxygen consumption and oxygen extraction | 75 min minus baseline
  Oxygen consumption: Renal blood flow multiplied by arterial-renal venous oxygen difference.
  Oxygen extraction: Ratio of renal oxygen consumption to renal oxygen delivery
Change in filtration fraction | 75 min minus baseline
  Ratio of glomerular filtration rate to renal plasma flow

CONTACTS AND LOCATIONS:
Overall Officials: Kristjan Karason, MD, PhD, Principal Investigator — Sahlgrenska University Hospital, Department of Cardiology
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Savarese G, Lund LH. Global Public Health Burden of Heart Failure. Card Fail Rev. 2017 Apr;3(1):7-11. doi: 10.15420/cfr.2016:25:2. PMID 28785469
- [Result] Hillege HL, Nitsch D, Pfeffer MA, Swedberg K, McMurray JJ, Yusuf S, Granger CB, Michelson EL, Ostergren J, Cornel JH, de Zeeuw D, Pocock S, van Veldhuisen DJ; Candesartan in Heart Failure: Assessment of Reduction in Mortality and Morbidity (CHARM) Investigators. Renal function as a predictor of outcome in a broad spectrum of patients with heart failure. Circulation. 2006 Feb 7;113(5):671-8. doi: 10.1161/CIRCULATIONAHA.105.580506. PMID 16461840
- [Result] Smith GL, Shlipak MG, Havranek EP, Masoudi FA, McClellan WM, Foody JM, Rathore SS, Krumholz HM. Race and renal impairment in heart failure: mortality in blacks versus whites. Circulation. 2005 Mar 15;111(10):1270-7. doi: 10.1161/01.CIR.0000158131.78881.D5. PMID 15769768
- [Result] Hillege HL, Girbes AR, de Kam PJ, Boomsma F, de Zeeuw D, Charlesworth A, Hampton JR, van Veldhuisen DJ. Renal function, neurohormonal activation, and survival in patients with chronic heart failure. Circulation. 2000 Jul 11;102(2):203-10. doi: 10.1161/01.cir.102.2.203. PMID 10889132
- [Derived] Lannemyr L, Ricksten SE, Rundqvist B, Andersson B, Bartfay SE, Ljungman C, Dahlberg P, Bergh N, Hjalmarsson C, Gilljam T, Bollano E, Karason K. Differential Effects of Levosimendan and Dobutamine on Glomerular Filtration Rate in Patients With Heart Failure and Renal Impairment:A Randomized Double-Blind Controlled Trial. J Am Heart Assoc. 2018 Aug 21;7(16):e008455. doi: 10.1161/JAHA.117.008455. PMID 30369310